CLINICAL TRIAL: NCT03359421
Title: Trauma Routing Algorithm for Pediatrics
Acronym: TRAP
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00047353
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Pediatric All; Trauma
Keywords: prehospital; aeromedical; trauma; ems; helicopter
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aeromedical transport: Patients transported to trauma center by helicopter
- Ground transport: Patients transported to trauma center by ground ambulance

SUMMARY:
Traumatic injury is the leading cause of pediatric death in the United States for those forty-four years of age and younger. Pediatric trauma patients generally have reduced mortality when treated at pediatric trauma centers rather than at adult centers or non-tertiary care facilities. However, nearly half the US pediatric population lives over fifty miles from a Level I or II Trauma Center. While air ambulances are readily available in many jurisdictions, few guidelines and little evidence dictate their appropriate use, especially with regard to pediatric trauma. Previous research is mixed regarding mortality benefit from helicopter Emergency Medical Services (EMS) in injured children. Previous attempts to develop appropriate field triage criteria have failed due to poor sensitivity and specificity for identifying the critically injured child. The current high rate of overtriage is particularly concerning in today's cost-conscious medical community. This research study aims to categorize pre-hospital pediatric trauma in North Carolina, to determine what benefits helicopter EMS provides in the North Carolina trauma system, and to formulate an enhanced screening tool for pre-hospital use to help determine which patients are suitable candidates for helicopter EMS transport.

DETAILED DESCRIPTION:
The North Carolina Trauma Registry will identify pediatric trauma patients between 0 and 18 years of age who presented directly to North Carolina Level 1 Trauma Centers from the field after sustaining injury from January 1st, 2013 and October 2017.

The analysis will be a retrospective cohort study by nature of the data set. Final methodology will be determined after Institutional Review Board approval and enlistment of statistical support through the Clinical and Translational Science Institute. Clinical and non-clinical factors will first be summarized with univariate analysis to provide a descriptive overview of the study population. These factors will include number of case-patients, demographics, scene address/location, time of injury, EMS agency involved, EMS call times, transport mechanism, time of transport, distance of transport, geographic area of injury, mechanism of injury, severity scores, Glasgow Coma Score, vital signs, receiving hospital name, and other variables. Similarly, interventions and outcomes will be compared between study groups through such factors such as length of emergency department stay, emergency department disposition, time to operating room, intubation status on arrival, administration of blood products, days of hospital stay, days of intensive care unit stay, days on ventilator, if viable organs were procured post-mortem, and mortality at given time points. Outcomes will be compared through regression analysis or related means.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric trauma victims 0-16 years old who are reported in the North Carolina Trauma Registry after presenting to a North Carolina Trauma Center between January 1st, 2013 and October, 2017.

Exclusion Criteria:

* Interfacility transport patients are excluded

Ages: 2 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients <16 years old involved in trauma that were transported to a North Carolina Trauma Center
Sampling Method: Probability Sample
Enrollment: 4801 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Survival | approximately 1 month or less
  Patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stopyra, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arfken CL, Shapiro MJ, Bessey PQ, Littenberg B. Effectiveness of helicopter versus ground ambulance services for interfacility transport. J Trauma. 1998 Oct;45(4):785-90. doi: 10.1097/00005373-199810000-00031. PMID 9783622
- [Background] Baxt WG, Moody P. The impact of a rotorcraft aeromedical emergency care service on trauma mortality. JAMA. 1983 Jun 10;249(22):3047-51. PMID 6854826
- [Background] Biewener A, Aschenbrenner U, Rammelt S, Grass R, Zwipp H. Impact of helicopter transport and hospital level on mortality of polytrauma patients. J Trauma. 2004 Jan;56(1):94-8. doi: 10.1097/01.TA.0000061883.92194.50. PMID 14749573
- [Background] Bledsoe BE, Wesley AK, Eckstein M, Dunn TM, O'Keefe MF. Helicopter scene transport of trauma patients with nonlife-threatening injuries: a meta-analysis. J Trauma. 2006 Jun;60(6):1257-65; discussion 1265-6. doi: 10.1097/01.ta.0000196489.19928.c0. PMID 16766969
- [Background] Chappell VL, Mileski WJ, Wolf SE, Gore DC. Impact of discontinuing a hospital-based air ambulance service on trauma patient outcomes. J Trauma. 2002 Mar;52(3):486-91. doi: 10.1097/00005373-200203000-00012. PMID 11901324
- [Background] Englum BR, Rialon KL, Kim J, Shapiro ML, Scarborough JE, Rice HE, Adibe OO, Tracy ET. Current use and outcomes of helicopter transport in pediatric trauma: a review of 18,291 transports. J Pediatr Surg. 2017 Jan;52(1):140-144. doi: 10.1016/j.jpedsurg.2016.10.030. Epub 2016 Oct 27. PMID 27852453
- [Background] Floccare DJ, Stuhlmiller DF, Braithwaite SA, Thomas SH, Madden JF, Hankins DG, Dhindsa H, Millin MG. Appropriate and safe utilization of helicopter emergency medical services: a joint position statement with resource document. Prehosp Emerg Care. 2013 Oct-Dec;17(4):521-5. doi: 10.3109/10903127.2013.804139. Epub 2013 Jul 8. PMID 23834231
- [Background] Lerner EB, Drendel AL, Cushman JT, Badawy M, Shah MN, Guse CE, Cooper A. Ability of the Physiologic Criteria of the Field Triage Guidelines to Identify Children Who Need the Resources of a Trauma Center. Prehosp Emerg Care. 2017 Mar-Apr;21(2):180-184. doi: 10.1080/10903127.2016.1233311. Epub 2016 Oct 6. PMID 27710155
- [Background] Michailidou M, Goldstein SD, Salazar J, Aboagye J, Stewart D, Efron D, Abdullah F, Haut ER. Helicopter overtriage in pediatric trauma. J Pediatr Surg. 2014 Nov;49(11):1673-7. doi: 10.1016/j.jpedsurg.2014.08.008. Epub 2014 Nov 6. PMID 25475816
- [Background] Mitchell AD, Tallon JM, Sealy B. Air versus ground transport of major trauma patients to a tertiary trauma centre: a province-wide comparison using TRISS analysis. Can J Surg. 2007 Apr;50(2):129-33. PMID 17550717
- [Background] Moront ML, Gotschall CS, Eichelberger MR. Helicopter transport of injured children: system effectiveness and triage criteria. J Pediatr Surg. 1996 Aug;31(8):1183-6; discussion 1187-8. doi: 10.1016/s0022-3468(96)90114-1. PMID 8863261
- [Background] Potoka DA, Schall LC, Gardner MJ, Stafford PW, Peitzman AB, Ford HR. Impact of pediatric trauma centers on mortality in a statewide system. J Trauma. 2000 Aug;49(2):237-45. doi: 10.1097/00005373-200008000-00009. PMID 10963534
- [Background] Sathya C, Alali AS, Wales PW, Scales DC, Karanicolas PJ, Burd RS, Nance ML, Xiong W, Nathens AB. Mortality Among Injured Children Treated at Different Trauma Center Types. JAMA Surg. 2015 Sep;150(9):874-81. doi: 10.1001/jamasurg.2015.1121. PMID 26106848
- [Background] Stewart CL, Metzger RR, Pyle L, Darmofal J, Scaife E, Moulton SL. Helicopter versus ground emergency medical services for the transportation of traumatically injured children. J Pediatr Surg. 2015 Feb;50(2):347-52. doi: 10.1016/j.jpedsurg.2014.09.040. Epub 2014 Oct 1. PMID 25638635
- [Background] Sullivent EE, Faul M, Wald MM. Reduced mortality in injured adults transported by helicopter emergency medical services. Prehosp Emerg Care. 2011 Jul-Sep;15(3):295-302. doi: 10.3109/10903127.2011.569849. Epub 2011 Apr 27. PMID 21524205
- [Background] Webman RB, Carter EA, Mittal S, Wang J, Sathya C, Nathens AB, Nance ML, Madigan D, Burd RS. Association Between Trauma Center Type and Mortality Among Injured Adolescent Patients. JAMA Pediatr. 2016 Aug 1;170(8):780-6. doi: 10.1001/jamapediatrics.2016.0805. PMID 27368110